CLINICAL TRIAL: NCT02866162
Title: Identification of the Molecular Bases of Syndromic Congenital Neutropenia With Development Anomalies
Brief Title: Screening for Genes in Patients With Congenital Neutropenia
Acronym: neutropenias
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Thauvin PARI 2013
Record Dates: First submitted 2016-08-05; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Congenital Neutropenia
MeSH Terms: conditions — Neutropenia, Severe Congenital, Autosomal Recessive 3

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- patients with neutropenia
  Interventions: Genetic: High-throughput exome sequencing

INTERVENTIONS:
Genetic: High-throughput exome sequencing

SUMMARY:
Syndromic congenital neutropenia (SCN) includes a heterogeneous group of diseases characterized by congenital neutropenia associated with the involvement of other organs. Most patients have syndromic congenital neutropenia, which does not correspond, either clinically or genetically, to any other previously described form. A large number of genes still have to be identified in these syndromic forms.

The aim of this study is to identify the molecular bases of congenital neutropenias that have not yet been classified, by taking advantage of high-throughput exome sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have provided written consent
* Patients with congenital neutropenia and mental retardation and/or a development anomaly (malformation, facial dysmorphism)
* Patients who accept a clinical evaluation, and to give at least one blood sample
* Screening for chromosomal microrearrangements by normal array-CGH

Exclusion Criteria:

* Persons without national health insurance cover
* Patients who do not meet the clinical and/or biological criteria
* Refusal to give written consent to take part in the study
* Refusal to give a blood sample
* Blood samples from parents not available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with syndromic congenital neutropenia with development anomalies
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Identification of a gene or genes responsible for congenital neutropenia syndromic | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France